CLINICAL TRIAL: NCT05900687
Title: Developing, Refining, and Testing a Mobile Health Question Prompt List in Gastroesophageal Reflux Disease
Brief Title: Developing and Testing Mobile Health Question Prompt List in Gastroesophageal Reflux Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Afrin Kamal, Clinical Assistant Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 62297
Record Dates: First submitted 2023-05-31; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-05

CONDITIONS: Gastroesophageal Reflux; Patient Activation
MeSH Terms: conditions — Gastroesophageal Reflux; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Focus Group (Aim 1) (No Intervention): Participants give feedback about day-to-day challenges with GERD.
- Focus Group (Aim 2) (No Intervention): Participants give feedback about mobile health app prototype
- mHealth app (Aim 3) (Experimental): Participants will be exposed to an app-based question prompt list with gamification features to promote medication adherence as part of their communication with their health provider.
  Interventions: Behavioral: Use of mHealth Question Prompt List app
- Standard of care (Aim 3) (No Intervention): Participants will be exposed to standard of care communication with their health provider (no mHealth app).

INTERVENTIONS:
Behavioral: Use of mHealth Question Prompt List app — mHealth Question Prompt List app that facilitates in asking questions with a physician during a consultation specific to GERD
  Other Names: Esophagus-Qs
  Arms: mHealth app (Aim 3)

SUMMARY:
More than 40% of patients with gastroesophageal reflux disease (GERD) experience uncontrolled, chronic symptoms. This proposal aims to improve symptom control for patients with GERD, by developing a mobile health (mHealth) Question Prompt List (QPL) intervention that helps patient ask questions with his/her physician about GERD. The first aim is to gather feedback about daily challenges of living with GERD. The second aim is to gather feedback on the prototype app. The third (primary) aim of this project is to develop the mHealth application and measure differences in patient activation when used compared to standard of care.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of GERD
* GerdQ score of >=8
* documented PPI use for GERD
* internet access at home or computer/mobile device
* ability to provide written or e-consent.

Exclusion Criteria:

* Established diagnosis that mimic GERD symptoms (e.g. achalasia by prior esophageal manometry)
* non-English speaking patients

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Patient Activation Measure Scale Score | month 3
  Patient Activation Measure is a measure of how much activation (knowledge and confidence) participants have in managing their health.
Patient Activation Measure Scale Score | month 6
  Patient Activation Measure is a measure of how much activation (knowledge and confidence) participants have in managing their health.

SECONDARY OUTCOMES:
Pill Count | months 3 and 6
  measures medication adherence
12-item Short Form Survey | months 3 and 6
  patient survey that measures health related quality of life
Gerd-Q | months 3 and 6
  patient survey that measures symptom severity of GERD

CONTACTS AND LOCATIONS:
Overall Officials: Afrin N Kamal, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No